CLINICAL TRIAL: NCT07099092
Title: Causal Mechanisms of Odor-Guided Behavior in Humans
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10002358; 002358-DA
Record Dates: First submitted 2025-07-31; First posted 2025-08-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-05

CONDITIONS: Normal Physiology
Keywords: Behavioral Tasks; Decision Making; fMRI; TUS

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment 1 (Experimental): TUS targeting PirC or sham TUS before olfactory perceptual decision making task
  Interventions: Device: TUS PirC; Device: TUS Sham
- Experiment 2 (Experimental): TUS targeting amygdala or sham TUS before olfactory conditioning task
  Interventions: Device: TUS Amy; Device: TUS Sham

INTERVENTIONS:
Device: TUS PirC — 120 seconds of 100 Hz low-intensity transcranial ultrasound stimulation targeting piriform cortex
  Arms: Experiment 1
Device: TUS Amy — 120 seconds of 100 Hz low-intensity transcranial ultrasound stimulation targeting amygdala
  Arms: Experiment 2
Device: TUS Sham — 120 seconds of 100 Hz low-intensity transcranial ultrasound stimulation targeting white matter

SUMMARY:
Background:

Little is known about how different regions of the brain responsible for the human sense of smell guide behaviors. In this study, researchers use a technique called transcranial ultrasound stimulation (TUS) to learn how odors affect the brain and behavior.

Objective:

To learn more about how the human sense of smell works.

Eligibility:

Healthy people aged 18 to 45 years who are right-handed.

Design:

Participants can volunteer for up to 2 different experiments. Each experiment requires 5 visits, each about 1 week apart. Food, alcohol, and caffeine may be limited before visits.

At the start of each visit, participants will answer questions about their health and how well they slept. Their sense of smell will be assessed.

Some visits may include tasks on a computer: While doing these tasks, participants may be asked to smell different odors, look at pictures, and listen to sounds. They will wear devices to track breathing, blood pressure, pulse, and other body responses to the tasks.

Some visits may include TUS: TUS uses ultrasound waves to briefly change brain activity. A gel will be applied to the scalp and hair, and a device will be placed against the participant s head. Participants may feel a tapping, pulling, and/or warm sensation on the skin underneath the device. They may also feel a twitch in their face, neck, arm, or leg muscles. Participants will do tasks before and after TUS.

Some visits will include functional magnetic resonance imaging (fMRI) scans. fMRI uses magnet and radio waves to capture images of the activity inside the brain. Participants will lie on a table that slides into a tube. They will perform tasks inside the scanner.

DETAILED DESCRIPTION:
Study Description:

Primary olfactory cortex has been implicated in a variety of odorguided behaviors in both animal models and humans. However, direct causal evidence for the functional role of different primary olfactory regions in humans is currently missing, due to the lack of non-invasive neuromodulation methods that can effectively target deep brain regions. With the recent advancement of transcranial focused ultrasound stimulation (TUS), this challenge can now be overcome. The goal of this protocol is to use TUS to temporarily modulate activity in primary olfactory cortex and thereby assess its contribution to olfactory function.

Objectives:

The primary objective is to determine the causal contribution of primary olfactory brain regions to olfactory functions. The secondary objective is to 1) evaluate the neural mechanisms by which these brain regions support these olfactory functions, and 2) assess the safety profile of TUS.

Endpoints:

The primary endpoint is to determine if TUS of olfactory cortices alters olfactory function. The secondary endpoints are to 1) evaluate whether TUS changes neural activity in olfactory regions and 2) assess the degree to which TUS elicits unwanted side effects in healthy adult participants.

ELIGIBILITY:
* INCLUSION CRITERIA

In order to be eligible to participate in this study, an individual must meet the following criteria:

1. Willingness to comply with all study procedures and availability for the duration of the study.
2. Aged 18-45 years old. Justification: Many neural processes change with age, and these changes could introduce unwanted variability in the measured signals.
3. In good general health based on the assessment of the Medical Advisory Investigator (MAI).
4. Agreement to adhere to Lifestyle Considerations throughout study duration. Consent signature will be documentation of meeting this criterion.
5. Right-handed.

EXCLUSION CRITERIA

Individuals who meet any of the following criteria will be excluded from participation:

1. Any neurological disorder that would increase seizure risk from TUS such as stroke, brain lesions, previous neurosurgery, epilepsy, any history of seizure or fainting episode of unknown cause, frequent severe headache, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than one month. The MAI will also retain discretion to exclude based on a history of a neurological illness or trauma that may compromise safety or data integrity.
2. Predisposition to seizures (e.g., first-degree family history of potentially hereditary epilepsy, etc.).
3. Current use (any use in the past week, daily use for more than one week within past 3 months) of any investigational drug or of any medications with psychotropic (e.g., benzodiazepines, etc.), or anti or pro-convulsive action. This will be determined at the discretion of the MAI.
4. Unable to undergo MRI, or TUS due to certain metallic or magnetic devices or implants in the body, claustrophobia, or other reasons.
5. History of noise-induced hearing loss or tinnitus.
6. Recent history (within past 12 months) of learning disability, major DSM-5 psychiatric disorder including major affective disorder, ADHD, obsessivecompulsive disorder, schizophrenia, or PTSD. This will be determined at the discretion of the MAI.
7. Pattern of alcohol and drug use in the past 12 months that is indicative of harmful use, loss of control over use, or physical dependence.
8. Daily nicotine, alcohol, or drug use (excluding caffeine) for at least 4 continuous weeks within the past 12 months.
9. Participation in any neuromodulation (e.g., TMS, TUS, tDCS, tACS, etc.) session (excluding the current protocol) in the past two weeks.
10. History of anaphylaxis, e.g., due to severe asthma, and/or food and non-food allergies (e.g., latex, detergents, soap, etc.).
11. History of significant chronic obstructive pulmonary disease (COPD) as increased levels of carbon dioxide may increase the susceptibility to cavitation and related tissue damage.
12. Uncorrected impairments in visual acuity severe enough to affect task participation.
13. Non-English speaking. Justification: Data integrity of some of the behavioral tasks used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing TUS and MRI procedures. The inability to effectively communicate TUS and MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants.
14. Serious skin disease or serious skin allergy on the hands or head. Justification: Gel will be applied to the skin on both head and hands, for transducer coupling and electrode placement, respectively. Allergic or adverse reactions to such treatment need to be ruled out.
15. Hyposmia, i.e., decreased sense of smell, or anosmia, i.e., loss of smell (Sniffin' Sticks Olfactory Identification Score < 10). Justification: The ability to smell is paramount to task performance.
16. Pregnancy. Justification: It is unknown whether MRI and pose risks to fetuses.
17. Any other condition that in the judgment of the investigators is incompatible with participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2035-07-14 (Estimated); Study Completion 2035-07-14 (Estimated)

PRIMARY OUTCOMES:
Task Performance<TAB> | Immediately after TUS
  Responses on behavioral tasks

SECONDARY OUTCOMES:
task-based fMRI | Immediately after TUS
  fMRI responses during behavioral task in Experiment 1
Report of symptoms | before, during and after TUS
  Report of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kahnt, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided